CLINICAL TRIAL: NCT03337620
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel 20 Week Study of the Efficacy and Safety of the Tx360® Nasal Applicator for Transnasal Sphenopalatine Ganglion Block in the Treatment of Chronic Migraine
Brief Title: Efficacy and Safety of Tx360® Transnasal Sphenopalatine Ganglion Block in the Treatment of Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tian Medical Inc. (Industry)
Collaborators: TAMM Net, Inc. (Unknown); Clinvest Research, LLC (Industry); Ki Health Partners. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-001TI
Record Dates: First submitted 2017-10-20; First posted 2017-11-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Headache, Migraine
Keywords: chronic
MeSH Terms: conditions — Migraine Disorders; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: multi-center, double blind, parallel, prospective, randomized; 28 days of screening; 4 weeks active treatment; 3 months of follow-up post-treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, investigator, study coordinator, and additional study staff will remain blinded. One member of the staff will assign subjects to a treatment group based on a computerized randomization number produced by a computer software system. The number will correspond to a kit number, of which the staff member will then use to prepare the Tx360® device for each of the subject's treatments during the 4-week treatment phase. If the clinical site has a pharmacy, it is preferred that the pharmacy receive the study medication and Tx360® devices, maintain custody of the study medication and Tx360® devices during the study, and prepared the medication in Tx360® devices for each subject's treatment, according to the computer-generated randomization. In order to maintain subject-blinding during the active phase of the study, subjects will be given a piece of lemon candy prior to each procedure as a taste distractor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bupivacaine (Active Comparator): Bupivacaine is a local anesthestic that will be delivered to the SPG by the Tx360 device.
  Interventions: Device: Tx360
- saline (Placebo Comparator): Saline is being used as a placebo treatment that will be delivered to the SPG by the Tx360 device.
  Interventions: Device: Tx360

INTERVENTIONS:
Device: Tx360 — Tx360 used to deliver active and placebo drug interventions to SPG.

SUMMARY:
This is a double blind placebo-controlled study which will evaluate the efficacy of bupivacaine compared to saline, delivered by the Tx360® device to the sphenopalatine ganglion (SPG), to treat chronic migraine headache. The Tx360® is a nasal applicator which is cleared through the FDA for transnasal medication delivery, including delivery to the SPG. The SPG has been implicated in a variety of cephalalgias. It is critical to the success of this intervention that the blocking agent be accurately delivered to this area as it is the only non-bony access to the pterygopalatine fossa (PPF). Subjects meeting inclusion/exclusion criteria will receive 12 intranasal treatments to the SPG over a period of 4 weeks with follow-up monthly for an additional 3 months post-treatment.

DETAILED DESCRIPTION:
This is a phase III, multi-center, randomized, double-blind, placebo-controlled, prospective, clinical trial examining the outcomes of subjects with chronic migraine headache who are treated with 0.3cc of 0.5% bupivacaine bilaterally vs 0.3cc of sterile water bilaterally, each delivered to the mucosal surface of the SPG through each nare with the Tx360® device.

Subjects must have a current history of ICHD-III beta migraine with > 14 headache days per month (with 8 or more being migraine) in the 3 months prior to the screening visit. Subjects will be required to have a stable history of doses of migraine prophylactic medication for at least 30 days prior to the start of the 28-day screening/baseline phase and for the duration of the study. At Visit 1, the subject will sign the informed consent indicating they are willing to participate in the study. Initially, subjects who meet the study criteria will participate in a 28-day screening/baseline phase. During the 28-day screening/baseline phase, all subjects will be monitored through the use of electronic Daily Headache Diary (DHD) to ensure they continue to meet all inclusion criteria, and none of the exclusion criteria.

If baseline criteria have been met at the end of the 28-day screening/baseline phase, the subject will return to the clinic for Visit 2 to be randomized into one of the two treatment groups and begin the 4-week treatment phase of the study. Subjects who meet all inclusion criteria, and none of the exclusion criteria, will be assigned to a treatment group based on a computerized randomization number produced by a computer software system. One hundred and eighty subjects will be randomized 1:1 to receive 0.3cc of 0.5% bupivacaine bilaterally or 0.3cc of sterile water bilaterally. One member of the staff will allocate study medication, based on the randomization plan, in a blinded fashion to subject, coordinator, and investigator. At Visit 2, the subject will receive the first treatment.

The subject will return to the clinic three times per week for treatments, totaling 12 treatments.

At visit 13, subjects will receive the last treatment and will be transitioned into the post-treatment phase of the study.

The subject will be followed for an additional 3 months during the post-treatment phase for a total of 20 weeks participation in the study. During this post-treatment phase, the subject will maintain the DHD at an 80% participation rate and two monthly phone visits will take place 1 and 2 months post treatment respectively.

The subject will complete the study at Visit 14 to the clinic for final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included that meet the following criteria:

  1. willing to participate and sign informed consent
  2. ability to understand informed consent and study procedures, including able to use the electronic Daily Headache Diary
  3. in general good health based on investigator's judgment
  4. male or female, age must be between 18 to 65 years of age, inclusive
  5. chronic migraine meeting the diagnostic criteria listed in the International Classification of Headache Disorders (ICHD-III beta version, 2013), as follows:

     1. History of frequent headaches suggestive of chronic migraine (at least 15 days per month with 8 or more being migraine) for at least three months prior to screening
     2. Verification of headache frequency through prospectively collected baseline information during the 28-day screening/baseline phase demonstrating headaches at least 15 days, with at least 8 days per month fulfilling any one of the following

        1. Qualify as being a migraine
        2. Relieved by migraine specific acute medications
  6. onset of migraine before age 50
  7. able to differentiate migraine from any other headache they may experience (e.g., tension-type headache)
  8. stable history of migraine at least 3 months prior to screening with headache free periods
  9. not currently taking a migraine preventive OR has been taking a stable dose of a preventive for at least 60 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period

     a) subjects on migraine preventative should have stable headache pattern
  10. subject is either not of childbearing potential, as defined in the methods section, or if they are of childbearing potential they agree either to remain abstinent or use (or have their partner use) an acceptable method of birth control for the duration of the study
  11. demonstrated compliance with the electronic Daily Headache Diary during the 28-day screening/baseline phase as defined by entry of headache data on a minimum of 22 to 28 days (80% diary compliance) in or completing the study.

Exclusion Criteria:

Subjects will be excluded that meet the following criteria:

1. unable to complete headache records (diary) as required by protocol
2. pregnant, actively trying to become pregnant, or breast-feeding
3. history of medication overuse (MO) of opioids, or butalbital, as defined by ICHD-III beta criteria in the previous 12 months and/or MO during 28-day screening/baseline phase (Appendix B).
4. history of hemiplegic migraine, basilar migraine, cervicogenic headache, occipital neuralgia or post-traumatic headache as defined by ICHD-III beta criteria (Post traumatic headache needs to have developed within 7 days of the following: injury to the head, regaining of consciousness following injury to the head, or discontinuation of medications that impair ability to send or report headache following the injury to the head.
5. has failed greater than 2 migraine preventative medications due to lack of efficacy after adequate trial
6. received onabotulinumtoxinA for migraine or for any medical or cosmetic reasons requiring injections in the head, face, or neck during the 4 months before screening.
7. has a planned military deployment within the 6 months post screening
8. has previously received SPG blocks using the Tx360®device
9. history of substance abuse and/or dependence within the past 5 years, in the judgment of the Investigator
10. unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure, in the judgment of the investigator
11. suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events, in the judgment of the investigator
12. any psychiatric condition with psychotic features, and/or any other psychiatric disorder not stable or well controlled, that would interfere in the ability to complete study activities
13. malignancy within the past year, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
14. nasal septal deformity such as cleft lip and palate, choanal atresia, atrophic rhinitis, rhinitis, or septal perforation
15. recent nasal/midface trauma (< 3 months)
16. nasal or facial fracture
17. recent nasal/sinus surgery (< 3 months)
18. bleeding disorder such as Von Willebrand disease or hemophilia
19. severe respiratory distress
20. neoplasm such as Angiofibroma, sinus tumor, granuloma
21. nasal congestion present more than 10 days with fever (temperature ≥ 100.4 F) and nasal mucous is an abnormal color
22. skin around and inside the nasal passage that is dry, cracked, oozing, or bleeding
23. recurrent nose bleeds
24. allergy to bupivacaine
25. has a score > 0 on question 9 of PHQ-9 at any visit
26. received any investigational agents within 30 days prior to Visit 1
27. plans to participate in another clinical study at any time during this study
28. have any other conditions that in the judgment of the Investigator would make the subject unsuitable for inclusion, or would interfere with the subject participating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Change in Number of Migraine Headaches During Treatment Phase | From 28-day screening/baseline phase to the end of the 4-week treatment phase.
  Evaluate the efficacy of bupivacaine delivered with the Tx360® device, based on the change in the number of migraine days during treatment.

SECONDARY OUTCOMES:
Change in Number of Migraine Headache Days Post-Treatment | From 28-day screening/baseline to end of one month post-treatment, end of two months post-treatment, and end of three months post treatments (EOS)
  Evaluate the efficacy of bupivacaine delivered with the Tx360® device, based on the change in the number of migraine days post-treatment.
Safety/Tolerability of TX360 Device Based on Adverse Effects | Measured per month from end of 28-day screening/baseline phase to end of the 4-week treatment phase, and end of one month post- treatment, end ot two months post-treatment, and end of 3 months post-treatment.(EOS)
  Evaluate the safety and tolerability of the Tx360® device in the prevention of chronic migraine based on reported adverse effects.

OTHER OUTCOMES:
Efficacy Evaluation Based on Change in Mean Headache Severity | Measured per month from end of 28-day screening/baseline phase to end of the 4-week treatment phase, and end of one month post- treatment, end ot two months post-treatment, and end of 3 months post-treatment.(EOS)
  Evaluate the efficacy of bupivacaine vs sterile water delivered with the Tx360® device, based on the change in the mean headache severity.
Efficacy Evaluation Based on Change in Mean Number of Headache Days per Month | Measured per month from end of 28-day screening/baseline phase to end of the 4-week treatment phase, and end of one month post- treatment, end ot two months post-treatment, and end of 3 months post-treatment.(EOS)
  Evaluate the efficacy of bupivacaine vs sterile water delivered with the Tx360® device, based on the change in the mean number of headache days per month.
Comparison of Response Rate | Measured per month from end of 28-day screening/baseline phase to end of the 4-week treatment phase, and end of one month post- treatment, end ot two months post-treatment, and end of 3 months post-treatment.(EOS)
  Compare the response rate of those in bupivacaine vs sterile water delivered with the Tx360® device.
Comparison of Acute Medication Required | Measured per month from end of 28-day screening/baseline phase to end of the 4-week treatment phase, and end of one month post- treatment, end ot two months post-treatment, and end of 3 months post-treatment.(EOS)
  Compare the need between treatment groups for acute medication based on number of doses of acute headache medication taken.
Evaluate Life Impact of Migraine Headaches | End of 28-day screening/baseline phase and end of 3 months post treatment.(EOS)
  Evaluate the impact of chronic migraine headaches on the subject's life (pain and disability) based on change in Migraine Disability Assessment (MIDAS) scores between treatment groups.
Evaluate Disease Management Impact on Change in PROMIS Score | Measured from end of 28-day screening/baseline phase and end of 3 months post treatment. (EOS) to end of treatment phase, and end of post treatment.
  Evaluate the subject's perceived impact of disease management based on change in Patient-Reported Outcomes Measurement Information System (PROMIS) scores between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tian Xia, MD, Study Chair — Tian Medical
Locations (11):
- United States (11):
  - Yale University, New Haven, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Crescent City Headache and Neurology Centre, Chalmette, Louisiana
  - MedVadis Research, Watertown, Massachusetts
  - Clinvest Research, LLC, Springfield, Missouri
  - Hudson Medical, New York, New York
  - North Suffolk Neurology, PC, Port Jefferson Station, New York
  - Womack Army Medical Senter, Fort Bragg, North Carolina
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Lone Star Neurology, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No